CLINICAL TRIAL: NCT04300491
Title: Monocentric Descriptive Study Focuses on the Feasibility, Safety and Benefits of Using a Specific Suspension Walking Device for Patients With Neurological Damage
Brief Title: Study Examines the Feasibility, Safety and Benefits of Using a Specific Suspension Walking Device for Patients With Neurological Damage
Acronym: Walk-Up
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0129
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Stroke; Traumatic Brain Injury; Incomplete Cervical Spinal Cord Injury; Other Brain Injuries
Keywords: Early mobilization; ICU; Brain injuries; Verticalization
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Beneficiaries of suspension walking
  Interventions: Other: Suspension walking training
- Non-Beneficiaries of suspension walking

INTERVENTIONS:
Other: Suspension walking training — Physiotherapy session, objective wlaking with body weight support using a specific device
  Groups: Beneficiaries of suspension walking

SUMMARY:
This monocentric descriptive study addresses feasibility, safety and benefits of using a specific suspension walking device for patients with severe neurological injuries in the neuroICU of Montpellier University Hospital, France. Analyzes are retrospective on data collected prospectively during standard practice. All adult neurological patients hospitalized for > 48 hours and requiring mechanical ventilation from January 2018 to January 2019 are included, and divided into two groups: beneficiaries of suspension walking during the ICU stay, and non-beneficiaries. Characteristics of the two groups are compared and reasons for not using suspension walking recorded (feasibility). After pooling all suspension walking sessions, changes in clinical parameters during sessions and occurrence of adverse events are described (tolerance).

DETAILED DESCRIPTION:
Background. Current literature and National guidelines recommend early mobilization in Intensive Care Units (ICU), including verticalization and walking. Verticalization for neurologic patients in ICU is challenging because of neurological impairments, risks of falls and of clinical worsening. In the neuroICU of Montpellier university hospital, France, a weight suspension system (LiteGait®) is used for gait training.

Objectives. To study the feasibility, safety and benefits of walking with the weight suspension system in a neuroICU. Feasibility involves the proportion of patients who benefited from suspension walking, reasons for not using it, physiotherapists' time required. Safety involves rate and causes of adverse events, changes in vital parameters and in pain. Benefits of suspension walking involves difference between delay for first suspension walking session and first walking session without suspension.

Design. Monocentric, descriptive study, using retrospective analyzes of prospectively-collected data during standard clinical and rehabilitation management in the neuroICU. It includes all adult neurological patients hospitalized for > 48 hours in the unit and requiring mechanical ventilation from January 2018 to January 2019. Exclusion criteria are death before sedation weaning; therapeutic limitation; complete spinal cord injury.

The study sample is divided into two groups: beneficiaries of suspension walking during the ICU stay, and non-beneficiaries. Criteria for using suspension walking used in standard practice in the unit are respiratory stability without mechanical ventilation (tracheostomy and/or oxygen therapy possible), hemodynamic and neurologic stability, sufficient respond to command (head control, ability to sit with aid, testing of one quadriceps > 3 or two quadriceps > 2).

Data collected include clinical description of patients upon ICU admission, duration of sedation, ventilation, hospitalization, and delay before first sitting on a chair, first walking without suspension. For beneficiaries of suspension walking, clinical status before session (pain, MRC testing, sitting balance, RASS, hemodynamic and respiratory parameters, medical equipment) and after session (pain, hemodynamic and respiratory parameters) are collected, as well as description of adverse events and consequences. For non-beneficiaries, reasons for not using suspension walking are collected.

Analyses will be mainly descriptive. Characteristics of beneficiaries and non-beneficiaries of suspension walking will be described and compared. Description of suspensi

ELIGIBILITY:
Inclusion criteria:

* Adults
* Severe Neurological injury
* Hospitalization > 48h in a unique Neuro-ICU
* Necessity of mechanical ventilation

Exclusion criteria:

* death before sedation weaning
* therapeutic limitation
* complete spinal cord injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Adults with Severe Neurological injury hospitalized in a unique Neuro-ICU from January 2018 to January 2019
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 1 day
  Number of adverse events assessed immediately during walking sessions

SECONDARY OUTCOMES:
pre-post session changes in pulse | 1 day
  pre-post session changes in pulse assessed immediately during walking sessions
oxygen saturation | 1 day
  oxygen saturation assessed immediately during walking sessions
blood pressure | 1 day
  blood pressure assessed immediately during walking sessions
Pain assessment | 1 day
  pain assessed immediately during walking sessions

CONTACTS AND LOCATIONS:
Overall Officials: claire Jourdan, MD.PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Jourdan C, Pradalier F, Chalard K, Ascher M, Miron Duran F, Pavillard F, Greco F, Mellouk M, Fournier S, Djanikian F, Laffont I, Gelis A, Perrigault PF. Body-weight support gait training in neurological intensive care: safety, feasibility, and delays before walking with or without suspension. J Neuroeng Rehabil. 2023 Dec 13;20(1):167. doi: 10.1186/s12984-023-01291-9. PMID 38093374